CLINICAL TRIAL: NCT03293394
Title: Rehabilitative Trial With Transcranial Direct Current Stimulation (tDCS) in Amyotrophic Lateral Sclerosis
Brief Title: Rehabilitative Trial With tDCS in Amyotrophic Lateral Sclerosis
Acronym: tDCS_MND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NP2743
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Results first posted 2019-11-22 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): 10 days anodal bilateral motor cortex and cathodal spinal tDCS
  Interventions: Device: Anodal bilateral motor cortex and cathodal spinal tDCS
- Sham tDCS (Placebo Comparator): 10 days sham bilateral motor cortex and sham spinal tDCS
  Interventions: Device: Sham bilateral motor cortex and sham spinal tDCS

INTERVENTIONS:
Device: Anodal bilateral motor cortex and cathodal spinal tDCS — 10 sessions of anodal bilateral motor cortex and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Real tDCS
Device: Sham bilateral motor cortex and sham spinal tDCS — 10 sessions of sham bilateral motor cortex and sham spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Sham tDCS

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a motor neuron disease, which is a group of neurological disorders that selectively affect motor neurons, the cells that control voluntary muscles of the body. The disorder causes muscle weakness and atrophy throughout the body due to the degeneration of the upper and lower motor neurons. Current drugs approved for ALS treatment only modestly slow disease progression.

Transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebral excitability in several neurodegenerative disorders and modulate intracortical connectivity measures.

In this randomized, double-blind, sham-controlled study, the investigators will evaluate whether a two-weeks' treatment with bilateral motor cortex anodal tDCS and spinal cathodal tDCS can improve symptoms in patients with amyotrophic lateral sclerosis and modulate intracortical connectivity, at short and long term.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a motor neuron disease, which is a group of neurological disorders that selectively affect motor neurons, the cells that control voluntary muscles of the body. The disorder causes muscle weakness and atrophy throughout the body due to the degeneration of the upper and lower motor neurons. Current drugs approved for ALS treatment only modestly slow disease progression.

Transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebral excitability in several neurodegenerative disorders and modulate intracortical connectivity measures.

In this randomized, double-blind, sham-controlled study, the investigators will evaluate whether a two-weeks' treatment with bilateral motor cortex anodal tDCS and spinal cathodal tDCS can improve symptoms in patients with amyotrophic lateral sclerosis and modulate intracortical connectivity, at short and long term.

Subjects will be randomized in two groups, one receiving a 10 day (5 days/week for 2 weeks) treatment with anodal bilateral motor cortex tDCS and cathodal spinal tDCS and the other receiving sham stimulation with identical parameters. After the intervention, patients will be reassessed with a clinical and neurophysiological evaluation at 2 weeks, 2 months and 6 months after treatment. Furthermore, blood neurofilaments will be measured at each time point.

Clinical evaluation will include the ALSFRS-R, ALSAQ-40, CBI, EQ-5D-5L, muscle strength evaluated with the MRC scale.

Neurophysiological evaluation will include measures of intracortical connectivity, evaluated with transcranial magnetic stimulation (TMS) as short interval intracortical inhibition (SICI-ICF), long interval intracortical inhibition (LICI), short interval intracortical facilitation (SICF).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of probable, laboratory-supported probable, or definite amyotrophic lateral sclerosis according to the El Escorial revised criteria
* Disease duration ≤ 24 months
* Disease progression in the past 3 months
* Score ≥ 2 at the item "swallowing" of the ALS Functional Rating Scale Revised
* Score ≥ 2 at the item "walking" of the ALS Functional Rating Scale Revised
* Treatment with steady regimen of riluzole for a minimum of 1 month before study entry, and desiring its continuation
* Able to give informed consent
* Written informed consent

Exclusion Criteria:

* Motor neuron diseases other than ALS
* Severe head trauma in the past
* History of seizures
* History of ischemic stroke or hemorrhage
* Pacemaker
* Metal implants in the head/neck region
* Severe comorbidity
* Intake of illegal drugs
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia; Alberto Benussi, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- AO Spedali Civili, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quartarone A, Lang N, Rizzo V, Bagnato S, Morgante F, Sant'angelo A, Crupi D, Battaglia F, Messina C, Girlanda P. Motor cortex abnormalities in amyotrophic lateral sclerosis with transcranial direct-current stimulation. Muscle Nerve. 2007 May;35(5):620-4. doi: 10.1002/mus.20737. PMID 17221883
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Menon P, Geevasinga N, Yiannikas C, Howells J, Kiernan MC, Vucic S. Sensitivity and specificity of threshold tracking transcranial magnetic stimulation for diagnosis of amyotrophic lateral sclerosis: a prospective study. Lancet Neurol. 2015 May;14(5):478-84. doi: 10.1016/S1474-4422(15)00014-9. Epub 2015 Apr 3. PMID 25843898
- [Background] Burrell JR, Kiernan MC, Vucic S, Hodges JR. Motor neuron dysfunction in frontotemporal dementia. Brain. 2011 Sep;134(Pt 9):2582-94. doi: 10.1093/brain/awr195. Epub 2011 Aug 11. PMID 21840887

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (2 Weeks)
Arm/Group | Real tDCS | Sham tDCS
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0
Period: Follow-up (6 Months)
Arm/Group | Real tDCS | Sham tDCS
Started | 20 | 10
Completed | 16 | 8
Not Completed | 4 | 2
Not completed — Adverse Event | 4 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis are reported for 30 participants who completed the first intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.9) | 63.9 (11.3) | 61.7 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 13 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 10 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 10 | 30
Disease Duration [Mean (Standard Deviation); unit: years] | 2.1 (1.4) | 1.8 (1.0) | 2.0 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Strength From Baseline
Description: A megascore is obtained by summing scores of single muscles (shoulder abductors, elbow flexors and extensors, wrist flexors, thumb opponent, hip flexors, knee flexors and extensors, and ankle dorsiflexors and extensors on both sides) manually evaluated according to the Medical Research Council (MRC) scale, which ranges from 0 (no movement) to 5 (normal contraction).
  The score for each muscle is summed, with scores ranging from 100 (no impairment) to 0 (most severe impairment).
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 74.7 (0.0) | 74.7 (0.0)
  2 Weeks | 76.4 (0.2) | 74.5 (0.3)
  2 Months | 76.4 (0.4) | 72.9 (0.6)
  6 Months | 75.9 (0.6) | 72.0 (0.9)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.001, ANCOVA

2. Secondary Outcome: Change in Short-interval Intracortical Inhibition (SICI) From Baseline
Description: By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of tDCS on short-interval intracortical inhibition (SICI) from baseline
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
millivolts
  Baseline | 1.0 (0.1) | 1.0 (0.1)
  2 weeks | 0.4 (0.1) | 1.0 (0.1)
  2 Months | 0.5 (0.1) | 0.9 (0.1)
  6 Months | 0.6 (0.1) | 1.0 (0.1)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.011, ANOVA

3. Secondary Outcome: Change in the ALSFRS-R Score From Baseline
Description: Change in the ALS Functional Rating Scale (ALSFRS-R) score from baseline. The ALSFRS provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The ALSFRS includes ten questions that rate the patients level of functional impairment in performing one of ten common tasks. Each task is rated on a five-point scale from 0 (can't do) to 4 (normal ability). Individual item scores are summed to produce a reported score of between 40 (no impairment) and 0 (severe impairment).
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
units on a scale
  Baselin | 31.5 (0.0) | 31.5 (0.0)
  2 Weeks | 32.5 (0.2) | 31.8 (0.3)
  2 Months | 32.0 (0.4) | 30.4 (0.5)
  6 Months | 30.4 (0.5) | 29.7 (0.7)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.190, ANCOVA

4. Secondary Outcome: Change of Quality of Life From Baseline: ALSAQ-40 Scale
Description: Change of quality of life from baseline evaluated with the ALSAQ-40 scale. The Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ) is a patient self-report health status scale. The ALSAQ is specifically used to measure the subjective well-being of patients with amyotrophic lateral sclerosis. There are 40 items/questions with 5 discrete scales: physical mobility (10 items), activities of daily living and independence (10 items), eating and drinking (3 items), communication (7 items), emotional reactions (10 items). Patients are asked to think about the difficulties they may have experienced during the last two weeks (e.g. I have found it difficult to feed myself). Patients are asked to indicate the frequency of each event by selecting one of 5 options (Likert scale):
  never/rarely/sometimes/often/always or cannot do at all. The total ranges from 0 (no impairment) to 160 (severe impairment).
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 45.0 (0.0) | 45.0 (0.0)
  2 Weeks | 40.1 (2.0) | 38.3 (2.8)
  2 Months | 38.8 (1.8) | 41.0 (2.5)
  6 Months | 41.9 (2.2) | 42.4 (3.1)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.652, ANCOVA

5. Secondary Outcome: Change of Quality of Life From Baseline: EQ-5D-5L Scale
Description: Change of quality of life from baseline evaluated with the EQ-5D-5L scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The scale ranges from 5 (no impairment) to 25 (severe impairment).
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 13.0 (0.0) | 13.0 (0.0)
  2 Weeks | 12.2 (0.5) | 13.6 (0.8)
  2 Months | 12.6 (0.5) | 14.2 (0.7)
  6 Months | 13.3 (0.6) | 14.3 (0.9)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.190, ANCOVA

6. Secondary Outcome: Change of Quality of Life From Baseline: EQ-VAS Scale
Description: Change of quality of life from baseline evaluated with the EQ-VAS scale. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. The scale ranges from 0 (severe impairment) to 100 (no impairment).
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 51.6 (0.0) | 51.6 (0.0)
  2 Weeks | 56.3 (2.0) | 46.1 (2.8)
  2 Months | 53.2 (2.2) | 42.7 (3.1)
  6 Months | 54.7 (2.9) | 40.2 (4.0)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.011, ANCOVA

7. Secondary Outcome: Change in Caregiver Burden (CBI)
Description: Change of quality of life from baseline evaluated with the CBI scale. The CBI scale is 24- item scale designed to assess the experience of caregivers of older people. The multidimensional instrument assesses five domains of burden (time-dependence, developmental, physical, social, and emotional). Items are scored on a 4-point scale, ranging from "not at all descriptive" to "very descriptive". The scale ranges from 0 (no impairment) to 96 (severe impairment).
Time Frame: Baseline - 2 weeks - 2 months - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 26.7 (0.0) | 26.7 (0.0)
  2 Weeks | 21.6 (1.1) | 30.0 (1.5)
  2 Months | 24.0 (1.4) | 30.4 (1.9)
  6 Months | 24.8 (1.3) | 30.7 (1.9)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.003, ANCOVA

8. Secondary Outcome: Change Intracortical Facilitation (ICF) From Baseline
Description: By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of tDCS on intracortical facilitation (ICF) from baseline
Time Frame: Baseline - 2 weeks - 2 month - 6 months
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 10
millivolts
  Baselin | 1.8 (0.1) | 1.7 (0.1)
  2 Weeks | 1.3 (0.0) | 1.7 (0.1)
  2 Months | 1.4 (0.1) | 1.7 (0.1)
  6 Months | 1.6 (0.0) | 1.6 (0.1)
Statistical Analysis 1: Comparison: Real tDCS vs Sham tDCS; Test type: Superiority; p = 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 6 Months follow-up
Description: Adverse event has been defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Real tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/20 | 2/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS (N=20) | Sham tDCS (N=10)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Worsening of Global Clinical Conditions (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03293394/Prot_SAP_000.pdf